CLINICAL TRIAL: NCT05096182
Title: Long-term Follow-up of Patients With Chronic Kidney Disease Who Had Administered Cellgram-CKD in PMC-P-12 Study
Status: Active, not recruiting | Type: Observational
Sponsor: Pharmicell Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: PMC-P-12-01
Record Dates: First submitted 2021-10-15; First posted 2021-10-27 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Renal Insufficiency, Chronic
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This long-term follow-up study is a 5-year long-term follow-up study to evaluate long-term safety in Cellgram-CKD subjects. (refer to ClinicalTrials.gov.Identifier: NCT05042206).

DETAILED DESCRIPTION:
This long-term follow-up study is a 5-year long-term follow-up study to evaluate long-term safety in Cellgram-CKD subjects. (refer to ClinicalTrials.gov.Identifier: NCT05042206).

The long-term safety of Cellgram-CKD is evaluated by monitoring whether or not an adverse event of special interest (AESI) occurs for 5 years from the date of administration in Cellgram-CKD subjects who voluntarily consented in writing to participate in the long-term follow-up study.

ELIGIBILITY:
Inclusion Criteria:

* Those who participated in the PMC-P-12 clinical trial and received Cellgram-CKD
* Subjects who consented in writing to this long-term follow-up study

Exclusion Criteria:

* Not Applicable

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic kidney disease who participated in the PMC-P-12 clinical trial, among those who received Cellgram-CKD, those who agreed to participate in this long-term follow-up study
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Observe the occurrence of Adverse Event of Special Interest (AESI). | 5 years from the date of administration of Cellgram-CKD
  AESI stands for Serious Adverse Event as follows.
  1. death
  2. Creation of neoplasms or malignancies in tissues or organs
  3. The development of an immune response, including the exacerbation or new development of a previous autoimmune disease
  4. Occurrence of Other delayed adverse events related to stem cell therapy

CONTACTS AND LOCATIONS:
Overall Officials: Hyosang Kim, Principal Investigator — Asan Medical Center Hospital
Locations (1):
- Asan Medical Center Hospital, Seoul, South Korea